CLINICAL TRIAL: NCT05868902
Title: A Registry of Cardiac PET and CardioFlux Magnetocardiography in Patients With Suspected Coronary Ischemia.
Acronym: Magneto-PET
Status: Recruiting | Type: Observational
Sponsor: Genetesis Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 1000-8
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Coronary; Ischemic
Keywords: Magnetocardiography; Coronary Ischemia
MeSH Terms: conditions — Ischemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Negative Cardiac PET: Participants without clinical significant findings for coronary ischemia on cardiac PET scan.
  Interventions: Device: CardioFlux Magnetocardiography
- Positive Cardiac PET: Participants with findings indicative of coronary ischemia on cardiac PET scan.
  Interventions: Device: CardioFlux Magnetocardiography

INTERVENTIONS:
Device: CardioFlux Magnetocardiography — The device is a magnetocardiography (MCG) scanner named CardioFlux, which is paired with a cloud processing software. CardioFlux devices are owned by Genetesis and are currently cleared for the acquisition, display, and analysis of magnetic fields generated by cardiac electrical activity (K182571, FDA clearance letter available for download online)

SUMMARY:
A multicenter observational data development registry collecting diagnostic measures via standard of care (SOC) cardiac PET in order gain a better understanding of how CardioFlux MCG may be used in the detection of coronary ischemia.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide informed consent
* Male or female, aged 40 and up (inclusive) at the time of enrollment
* Clinical suspicion of myocardial ischemia that clinician desired cardiac PET
* Completed cardiac PET within 2 weeks prior to study enrollment

Exclusion Criteria:

* Patients unable to fit into CardioFlux device.
* Patients unable to lie supine for 5 minutes.
* Patients with implanted ferromagnetic objects above the costal margin of the rib cage (implanted pacemakers, cardioverter/defibrillators, infusion pumps, and/or neuro stimulators). NOTE: Sternotomy wires stents are acceptable
* Ongoing atrial fibrillation or atrial flutter
* Life expectancy <1 yrs. due to non-cardiovascular comorbidity

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women age 40 and up with suspected or confirmed coronary ischemia who are scheduled to undergo diagnostic cardiac PET, for non-emergent diagnostic purposes at an enrolling clinical trial center.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-08-28 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To collect diagnostic data using SOC diagnostic cardiac PET testing for the purposes of gaining a better understanding of how CardioFlux MCG may be used in the detection of coronary ischemia | 24 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cleveland Clinic, Cleveland, Ohio
  - Kettering Health, Kettering, Ohio

IPD SHARING:
Plan to Share IPD: No